CLINICAL TRIAL: NCT02203643
Title: A MULTICENTER, RANDOMIZED, OPEN LABEL PHASE II STUDY OF CARFILZOMIB, CYCLOPHOSPHAMIDE AND DEXAMETHASONE (CCyd) as Pre Transplant INDUCTION and Post Transplant Consolidation or CARFILZOMIB, LENALIDOMIDE AND DEXAMETHASONE (CRd) as Pre Transplant INDUCTION and Post Transplant Consolidation or Continuous Treatment With CARFILZOMIB, LENALIDOMIDE AND DEXAMETHASONE (12 Cycles) Without Transplant, All Followed by MAINTENANCE With LENALIDOMIDE (R) Versus LENALIDOMIDE AND CARFILZOMIB (CR) IN NEWLY DIAGNOSED MULTIPLE MYELOMA (MM) PATIENTS ELEGIBLE FOR AUTOLOGOUS TRANSPLANT
Brief Title: Evaluation of the Safety and the Efficacy of Carfilzomib Combined With Cyclophosphamide and Dexamethasone (CCyd) or Lenalidomide and Dex (CRd) Followed by ASCT or 12 Cycles of Carf Combined With Dex and Len for Patients Eligible for ASCT With Newly Diagnosed Multiple Myeloma.
Acronym: FORTE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mario Boccadoro (Other)
Responsible Party: Sponsor-Investigator, Mario Boccadoro, MD, University of Turin, Italy
Organization: University of Turin, Italy (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UNITO-MM-01 / FORTE
Record Dates: First submitted 2014-06-30; First posted 2014-07-30 (Estimated); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: MULTIPLE MYELOMA (MM)
MeSH Terms: conditions — Multiple Myeloma | interventions — carfilzomib; Cyclophosphamide; Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- CCyd (Experimental): Carfilzomib Cyclophosphamide and Dexamethasone administered for 4 28-day cycles. This treatment will be followed by autologous stem cell transplantation (ASCT). Carfilzomib Cyclophosphamide and Dexamethasone administered for 4 28-day cycles, as consolidation treatment.
  After the end of consolidation all patients will be randomized to receive:
  Lenalidomide or Lenalidomide and Carfilzomib until any sign of progression or intolerance.
  Interventions: Drug: Carfilzomib; Drug: Cyclophosphamide; Drug: Dexamethasone
- CRd (Experimental): Carfilzomib Lenalidomide and Dexamethasone administered for 4 28-day cycles. This treatment will be followed by autologous stem cell transplantation (ASCT). Carfilzomib Cyclophosphamide and Dexamethasone administered for 4 28-day cycles, as consolidation treatment.
  After the end of consolidation all patients will be randomized to receive:
  Lenalidomide or Lenalidomide and Carfilzomib until any sign of progression or intolerance.
  Interventions: Drug: Carfilzomib; Drug: Lenalidomide; Drug: Dexamethasone
- CRd long treatment (Experimental): Carfilzomib Lenalidomide and Dexamethasone administered for 4 28-day cycles. Stem cells collection will be performed. Carfilzomib Lenalidomide and Dexamethasone administered for 8 28-day cycles.
  After that all patients will be randomized to receive:
  Lenalidomide or Lenalidomide and Carfilzomib until any sign of progression or intolerance.
  Interventions: Drug: Carfilzomib; Drug: Lenalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Carfilzomib
Drug: Cyclophosphamide
  Arms: CCyd
Drug: Lenalidomide
  Other Names: Revlimid
  Arms: CRd; CRd long treatment
Drug: Dexamethasone

SUMMARY:
This study will evaluate the safety and the efficacy of carfilzomib combined with cyclophosphamide and dexamethasone (CCyd) or lenalidomide and dexamethasone (CRd) followed by autologous transplantation ASCT or 12 cycles of carfilzomib combined with dexamethasone and lenalidomide for patients eligible for ASCT with newly diagnosed multiple myeloma. As a secondary endpoint this study will evaluate the best maintenance treatment between lenalidomide and lenalidomide combined with carfilzomib.

Four hundred seventy-seven patients, males and females aged > 18 years, enrolled in several sites, will take part in this study.

The duration of the study is approximately 5 years.

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 18 years Newly diagnosed MM based on standard CRAB criteria (see appendix B). Patient < 65 years eligible for ASCT. Patient has measurable disease according to IMWG (International Myeloma Working Group) criteria.

Patient has given voluntary written informed consent. Patient agrees to use acceptable methods for contraception. Patient has a Karnofsky performance status ≥ 60%

Pretreatment clinical laboratory values within 30 days of enrolment:

Platelet count ≥50 x 109/L (≥30 x 109 /L if myeloma involvement in the bone marrow is > 50%) Absolute neutrophil count (ANC) ≥ 1 x 109/L without the use of growth factors Corrected serum calcium ≤14 mg/dL (3.5 mmol/L) Alanine transaminase (ALT): ≤ 3 x the Upper Limit Normal (ULN) Total bilirubin: ≤ 2 x the ULN Calculated or measured creatinine clearance: ≥ 30 mL/minute. LVEF≥40%. 2-D transthoracic echocardiogram (ECHO) is the preferred method of evaluation. Multigated Acquisition Scan (MUGA) is acceptable if ECHO is not available Life expectancy ≥ 3 months

Exclusion Criteria:

Previous treatment with anti-myeloma therapy (does not include radiotherapy, bisphosphonates, or a single short course of steroid < to the equivalent of dexamethasone 40 mg/day for 4 days) Patients with non-secretory MM unless serum free-light chains are present and the ratio is abnormal or a plasmocytoma with minimum largest diameters of > 2 cm Patients ineligible for autologous transplantation Pregnant or lactating females

Presence of:

Clinical active infectious hepatitis type A, B, C or HIV Acute active infection requiring antibiotics or infiltrative pulmonary disease Myocardial infarction or unstable angina ≤ 4 months or other clinically significant heart disease Peripheral neuropathy or neuropathic pain grade 2 or higher, as defined by National Cancer Institute Common Toxicity Criteria (NCI CTC) 4.0 Known history of allergy to Captisol ® (a cyclodextrin derivative used to solubilize carfilzomib) Contraindication to any of the required drugs or supportive treatments Invasive malignancy within the past 3 years Serious medical condition, laboratory abnormality or psychiatric illness that prevented the subject from the enrolment or place the subject at unacceptable risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 477 (Actual)
Dates: Start 2015-02; Primary Completion 2016-10 (Actual); Study Completion 2026-03-26 (Estimated)

PRIMARY OUTCOMES:
Efficacy in term of at least Very Good Partial Response (VGPR) | Up to 2 years
  The efficacy, in term of at least VGPR, of the combination of carfilzomib, dexamethasone with cyclophosphamide or lenalidomide after 4 cycles of induction treatment in newly diagnosed MM patients eligible for ASCT.

SECONDARY OUTCOMES:
sCR rate | up to 1 year
  the stringent complete response (sCR) rate in the 3 arms after complete primary therapy (induction, ASCT and consolidation for the transplant arms and after 12 cycles in the long treatment arm) in an explorative manner.
Safety as incidence of grade 3/4 adverse events | Up to 3 years
  the safety in the 3 induction/consolidation arms and in the 2 maintenance arms.
Survival | Up to 5 years
  the survival in the 3 induction/consolidation arms and in the 2 maintenance arms.
Correlation between tumor response and outcome with baseline prognostic factors. | up to 5 years
Minimal Residual Disease (MRD) | up to 5 years
  Minimal Residual Disease
Survival after relapse | up to 7 years
  the survival after relapse

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Palumbo, MD, Principal Investigator — University of Turin, Italy
Locations (1):
- IRCCS--CROB --CROB di Rionero in di Rionero in Vulture, Rionero in Vulture, Italy

REFERENCES:
- [Derived] D'Agostino M, Rota-Scalabrini D, Belotti A, Bertamini L, Arigoni M, De Sabbata G, Pietrantuono G, Pascarella A, Tosi P, Pisani F, Pescosta N, Ruggeri M, Rogers J, Olivero M, Garzia M, Galieni P, Annibali O, Monaco F, Liberati AM, Palmieri S, Stefanoni P, Zamagni E, Bruno B, Calogero RA, Boccadoro M, Musto P, Gay F. Additional copies of 1q negatively impact the outcome of multiple myeloma patients and induce transcriptomic deregulation in malignant plasma cells. Blood Cancer J. 2024 Jun 7;14(1):94. doi: 10.1038/s41408-024-01075-x. PMID 38849344
- [Derived] D'Agostino M, Bertuglia G, Rota-Scalabrini D, Belotti A, More S, Corradini P, Oliva S, Ledda A, Grasso M, Pavone V, Ronconi S, Vincelli ID, Ballanti S, Velluti C, Cellini C, Gozzetti A, Palmas AD, Gamberi B, Mancuso K, Paris L, Zambello R, Petrucci MT, Bruno B, Musto P, Gay F. Predictors of unsustained measurable residual disease negativity in patients with multiple myeloma. Blood. 2024 Feb 15;143(7):592-596. doi: 10.1182/blood.2023022080. PMID 38048557
- [Derived] Mina R, Musto P, Rota-Scalabrini D, Paris L, Gamberi B, Palmas A, Aquino S, de Fabritiis P, Giuliani N, De Rosa L, Gozzetti A, Cellini C, Bertamini L, Capra A, Oddolo D, Vincelli ID, Ronconi S, Pavone V, Pescosta N, Cea M, Fioritoni F, Ballanti S, Grasso M, Zamagni E, Belotti A, Boccadoro M, Gay F. Carfilzomib induction, consolidation, and maintenance with or without autologous stem-cell transplantation in patients with newly diagnosed multiple myeloma: pre-planned cytogenetic subgroup analysis of the randomised, phase 2 FORTE trial. Lancet Oncol. 2023 Jan;24(1):64-76. doi: 10.1016/S1470-2045(22)00693-3. Epub 2022 Dec 14. PMID 36528035
- [Derived] Bertamini L, Oliva S, Rota-Scalabrini D, Paris L, More S, Corradini P, Ledda A, Gentile M, De Sabbata G, Pietrantuono G, Pascarella A, Tosi P, Curci P, Gilestro M, Capra A, Galieni P, Pisani F, Annibali O, Monaco F, Liberati AM, Palmieri S, Luppi M, Zambello R, Fazio F, Belotti A, Tacchetti P, Musto P, Boccadoro M, Gay F. High Levels of Circulating Tumor Plasma Cells as a Key Hallmark of Aggressive Disease in Transplant-Eligible Patients With Newly Diagnosed Multiple Myeloma. J Clin Oncol. 2022 Sep 20;40(27):3120-3131. doi: 10.1200/JCO.21.01393. Epub 2022 Jun 6. PMID 35666982
- [Derived] Gay F, Musto P, Rota-Scalabrini D, Bertamini L, Belotti A, Galli M, Offidani M, Zamagni E, Ledda A, Grasso M, Ballanti S, Spadano A, Cea M, Patriarca F, D'Agostino M, Capra A, Giuliani N, de Fabritiis P, Aquino S, Palmas A, Gamberi B, Zambello R, Petrucci MT, Corradini P, Cavo M, Boccadoro M. Carfilzomib with cyclophosphamide and dexamethasone or lenalidomide and dexamethasone plus autologous transplantation or carfilzomib plus lenalidomide and dexamethasone, followed by maintenance with carfilzomib plus lenalidomide or lenalidomide alone for patients with newly diagnosed multiple myeloma (FORTE): a randomised, open-label, phase 2 trial. Lancet Oncol. 2021 Dec;22(12):1705-1720. doi: 10.1016/S1470-2045(21)00535-0. Epub 2021 Nov 11. PMID 34774221